CLINICAL TRIAL: NCT06622369
Title: The Effect of Virtual Reality on Fear, Pain and Anxiety in Children Undergoing Circumcision: A Randomized Controlled Study
Brief Title: The Effect of Virtual Reality on Fear, Pain and Anxiety in Children Undergoing Circumcision
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Katip Celebi University (Other)
Responsible Party: Principal Investigator, ELİZ GECTAN, Principal Investigator, Izmir Katip Celebi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 1734
Record Dates: First submitted 2024-09-29; First posted 2024-10-02 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-09

CONDITIONS: Virtual Reality
Keywords: pain; anxiety; fear; virtual reality
MeSH Terms: conditions — Pain; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Randomised controlled study
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental;:Virtual Reality-Game group (Experimental): Virtual Reality-Game group Before the circumcision procedure, patients in the VR group will be given a 5-minute training including instructions for the use of the virtual reality. Children in the game group will be allowed to choose a game of their choice compatible with virtual reality. Children in this group will be allowed to play the game of their choice for 10-15 minutes before the procedure. VR will be disinfected before and after each use in terms of infection risk.
  Interventions: Other: Virtual Reality-Game group
- Experimental: Virtual Reality-Cartoon group (Experimental): Virtual Reality-Cartoon group Before the circumcision procedure, patients in the VR group will be given a 5-minute training including instructions for the use of the virtual reality. Children in the cartoon-video group will be allowed to choose a cartoon of their choice compatible with virtual reality. Children in this group will be allowed to watch the cartoon of their choice for 10-15 minutes before the procedure. VR will be disinfected before and after each use in terms of infection risk.
  Interventions: Other: Virtual Reality-Cartoon-video group
- No Intervention (No Intervention): Children in the control group will not be subjected to any distraction method. The routine procedure of the clinic will be applied.

INTERVENTIONS:
Other: Virtual Reality-Game group — Children in the play group will be allowed to choose a game that is compatible with virtual reality. Children in this group will be allowed to play the game they want for 10-15 minutes before the procedure. VR will be disinfected before and after each use
  Arms: Experimental;:Virtual Reality-Game group
Other: Virtual Reality-Cartoon-video group — Children in the cartoon-video group will be allowed to choose a cartoon they want compatible with virtual reality. Children in this group will be allowed to watch the cartoon they want for 10-15 minutes before the procedure. VR will be disinfected before and after each use in terms of infection risk.
  Arms: Experimental: Virtual Reality-Cartoon group

SUMMARY:
The aim of this study is to investigate the effect of virtual reality and cartoons and games on the anxiety, fear and post-procedural pain levels of children aged 7-12 years who will undergo circumcision. The population of the study will consist of children aged 7-12 years who are planned to undergo circumcision in the pediatric urology clinic of İzmir Bakırçay University Çiğli and Training and Research Hospital between September 2024 and September 2025. The sample of the study will consist of children who meet the inclusion criteria on the specified dates and whose parents/legal guardians and themselves agree to participate in the study. Descriptive Characteristics Form, Vital Symptom Form, Child Fear Scale, Child Anxiety Scale-Disposition (CAS-D) and Child Fear Scale will be used to collect the data.

DETAILED DESCRIPTION:
Virtual Reality-Game group Before the circumcision procedure, patients in the VR group will be given a 5-minute training including instructions for the use of the virtual reality. Children in the game group will be allowed to choose a game compatible with virtual reality. Children in this group will be allowed to play the game of their choice for 10-15 minutes before the procedure. VR will be disinfected before and after each use in terms of infection risk.

Virtual Reality-Cartoons-Video group Before the circumcision procedure, patients in the VR group will be given a 5-minute training including instructions for the use of the virtual reality. Children in the cartoon-video group will be allowed to choose a cartoon of their choice compatible with virtual reality. Children in this group will be allowed to watch the cartoon of their choice for 10-15 minutes before the procedure. In terms of infection risk, VR will be disinfected before and after each use.

Control group Children in the control group will not be subjected to any distraction method. The routine procedure of the clinic will be applied.

Data Collection Phase 1: The study will start after ethics committee and institutional permissions are obtained. The researcher will inform the children and their parents about the study and the verbal and written consent of the participants will be obtained. Children who will undergo circumcision will be randomly assigned to the VR groups or the control group.

Phase 2: "Descriptive Characteristics Form", 'Child Fear Scale', 'Child Anxiety Scale-Conditionality (CAS-D)' will be completed for children in all groups before the circumcision procedure.

Phase 3: Children in the VR-game group will be asked to play a game of their choice for 10-15 minutes before the procedure. Children in the VR-cartoon-video group will be asked to watch a cartoon of their choice for 10-15 minutes.

Stage 4: Before the procedure, the physiologic parameters of the children in all groups will be recorded on the "Vital Signs Record Form".

5. After the procedure, "Child Fear Scale", "Child Anxiety Scale-Conditioning (CAS-D)" and "Visual Analog Scale" and "Life Findings Record Form" will be filled out for the children in all groups.

ELIGIBILITY:
Inclusion Criteria:

* Children between the ages of 7 and 12,
* The parent/legal guardian or the child himself/herself agrees to participate in the study
* Has not undergone any surgical operation before
* He was hospitalized for a circumcision
* No communication problems (visual, hearing, mental)

Exclusion Criteria:

* Chronic pain
* Eyeglass wear

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 105 (Estimated)
Dates: Start 2024-09-19 (Actual); Primary Completion 2025-09-19 (Estimated); Study Completion 2025-09-19 (Estimated)

PRIMARY OUTCOMES:
Fear assesed by Child Fear Scale | Procedure -Before the circumcision
  The Child Fear Scale (CFS), this one-item scale measures procedure-related fear in children, consists of five sex-neutral faces, ranges from 0 (no fear) to extreme fear.
Fear assesed by Child Fear Scale | Procedure -After the circumcision
  The Child Fear Scale (CFS), this one-item scale measures procedure-related fear in children, consists of five sex-neutral faces, ranges from 0 (no fear) to extreme fear.
Anxiety assesed by Children Anxiety Meter-State | Procedure -Before the circumcision
  The Children's Anxiety Meter (CAM-S). The Children's Anxiety Meter assesses children's anxiety and uses before medical procedures. This scale is drawn like a thermometer with a bulb at the bottom and also includes horizontal lines at intervals going up to the top (0-10).
Anxiety assesed by Children Anxiety Meter-State | Procedure -After the circumcision
  The Children's Anxiety Meter (CAM-S). The Children's Anxiety Meter assesses children's anxiety and uses before medical procedures. This scale is drawn like a thermometer with a bulb at the bottom and also includes horizontal lines at intervals going up to the top (0-10).
Visual Analog Scale | Procedure -After the circumcision
  The extremes of the line are 0 (no pain at all) and 10 (unbearable pain). In pain assessment with this scale, the child is asked to place a mark on a point between 0 and 10 to indicate the level of pain or to express it verbally

SECONDARY OUTCOMES:
Children's heart rate | Procedure -Before the circumcision
Children's heart rate | Procedure -After the circumcision
Children's respiratory rate | Procedure -Before the circumcision
Children's respiratory rate | Procedure -After the circumcision
Children's oxygen saturation | Procedure -Before the circumcision
Children's oxygen saturation | Procedure -After the circumcision

CONTACTS AND LOCATIONS:
Locations (1):
- Izmir Bakircay University Cigli Training and Research Hospital, Izmir, Turkey (Türkiye)